CLINICAL TRIAL: NCT05090956
Title: Mise au Point de Protocoles RMN Sur l'Imageur Philips 3T installé Sur le Site du Pavillon Baudot du CHU Purpan à Toulouse
Brief Title: Developpement of 3T MRI Protocol
Acronym: (MISAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C11-43; 2012-A00288-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-09-07; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Healthy; Adult ALL; MRI
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- control (Experimental): MRI exam; The sequences to be performed will be presented to the subject according to the focus to be performed. maximal duration of the exam: 2 hours (including subject set up)
  Interventions: Other: mri

INTERVENTIONS:
Other: mri

SUMMARY:
Since January 2010, a new magnetic resonance imaging scanner (Philips 3T, Achieva) is installed on the Baudot Building in Toulouse hospital. This tool, is completely dedicated to the research. It was installed with sequences RMN supplied by the manufacturer.

Imagers also contain an instrumentation susceptible to evolution and/or to adjustment (antennas radio frequency, sheath of gradients, elements of physiological monitoring (for example control of the breath), regulation of the homogeneity of the magnetic field).

This MRI scanner and this instrumentation are used for anatomical examinations or for paradigms of cognitiveresearch (for example of detection of intellectual activations following simple stimuli of fingers movement, visual tasks, or of mental processes).

The developpement of this equipment is going to favor the emergence of numerous projects and new themes, up to there adressed by other techniques (psychophysics, EEG).

To obtain good quality signals and know the practical limits of this imager, it is thus necessary that the researchers doctors, physicists and engineers, can finalize on volunteers' significant number, all the sequences RMN necessary for the use of these tools for the research.

These developments are going to get organized around four main axes:

1 the control of the geometrical distortions (generated by the introduction of an object within the magnetic field) 2 Optimization of the parameters of sequences to improve the contrast and the spatial resolution of the obtained images 3 the development of new sequences 4 the feasibility study of the protocols of functional MRI

ELIGIBILITY:
Inclusion Criteria:

Healthy adult, age = 18 years;

* Visual, hearing , oral or written capacities and expression sufficient for the suitable realization of the tests;
* Obtaining of the informed consent of the subject.

Exclusion Criteria:

* Subjects presenting a neurological, psychiatric history;
* Subjects under chronic medication which can influence the intellectual activity;
* Subjects presenting a contraindication to the MRI (carriers of a pacemaker, an implanted material(equipment) activated by an electric, magnetic or mechanical system, carriers of haemostatic clips of anévrysmes intracérébraux or carotid arteries, carriers of orthopaedic, claustrophobic implants);
* Subjects refusing to be informed about the possible presence of an anatomical anormality;
* administrative Problems: impossibility to give about the information, no insurance, refusal to sign the consent, under guardianship subject ;
* Subjects participating in another protocol • pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-06-08 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
quality of MRI images | 90 months
  assessment of distortion of MRI images

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm U825, Toulouse, France